CLINICAL TRIAL: NCT03209726
Title: Assessment of Subcutaneous Implantable Cardioverter Defibrillator Eligibility With 12-lead Electrocardiogram
Brief Title: Assessment of S-ICD Eligibility With 12-Lead ECG
Acronym: EL-SID
Status: Completed | Type: Observational
Sponsor: Larisa Tereshchenko (Other)
Responsible Party: Sponsor-Investigator, Larisa Tereshchenko, Associate Professor of Medicine, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Other Study IDs: STUDY00016034
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Implantable Defibrillator User

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to develop an approach to determine eligibility for subcutaneous ICD by analyzing routine clinical 12-lead electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* medical condition, predisposing patient to life-threatening ventricular arrhythmias, eligible for currently approved ICD indications for primary or secondary prevention of sudden cardiac death

Exclusion Criteria:

* Acute medical condition (e.g. acute myocardial infarction, severe trauma, post-surgery, admitted to ICU)
* End stage organ failure
* Pregnancy
* Patient, legal guardian or authorized representative is unable or unwilling to cooperate or give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ICD implantation for currently approved indications.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Amplitudes of R- and T-waves (and R/T ratios) on a special precordial ECG | at the day of ECG recording (cross-sectional study)
  Amplitudes of R- and T-waves (and R/T ratios) on a special ECG (recorded for Subcutaneous ICD eligibility assessment)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Thomas JA, Perez-Alday EA, Hamilton C, Kabir MM, Park EA, Tereshchenko LG. The utility of routine clinical 12-lead ECG in assessing eligibility for subcutaneous implantable cardioverter defibrillator. Comput Biol Med. 2018 Nov 1;102:242-250. doi: 10.1016/j.compbiomed.2018.05.002. Epub 2018 May 8. PMID 29754992
- [Result] Wang L, Javadekar N, Rajagopalan A, Rogovoy NM, Haq KT, Broberg CS, Tereshchenko LG. Eligibility for subcutaneous implantable cardioverter-defibrillator in congenital heart disease. Heart Rhythm. 2020 May;17(5 Pt B):860-869. doi: 10.1016/j.hrthm.2020.01.016. PMID 32354451